CLINICAL TRIAL: NCT00004256
Title: Randomised Phase II Study of GM-CSF to Reduce Severity of Mucositis Caused by Accelerated Radiotherapy of Laryngeal Cancer
Brief Title: Sargramostim to Prevent Mucositis in Patients Receiving Radiation Therapy for Laryngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000067503; RMNHS-GMCSF; EU-99041
Record Dates: First submitted 2000-01-28; First posted 2003-08-25 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2006-08

CONDITIONS: Head and Neck Cancer; Oral Complications; Radiation Toxicity
Keywords: stage I laryngeal cancer; stage II laryngeal cancer; recurrent laryngeal cancer; oral complications; radiation toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Laryngeal Neoplasms | interventions — sargramostim; Radiotherapy

INTERVENTIONS:
Biological: sargramostim
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as sargramostim may protect normal cells from the side effects of radiation therapy.

PURPOSE: Randomized phase II trial to determine the effectiveness of sargramostim in preventing mucositis in patients who are receiving radiation therapy for laryngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sargramostim (GM-CSF) in reducing the duration and severity of mucositis resulting from accelerated radiotherapy in patients with laryngeal carcinoma.
* Determine the effect of GM-CSF on quality of life aspects of these patients as assessed by nutritional status, analgesic use, and days in the hospital.

OUTLINE: This is a randomized study.

Patients receive radiotherapy in 16 fractions over 21 days. Patients are randomly allocated to one of two treatment arms before scheduled radiotherapy begins.

* Arm I: Patients receive sargramostim (GM-CSF) SC daily for 14 days beginning on day 14 of the course of radiotherapy.
* Arm II: Patients do not receive GM-CSF. Patients are followed weekly until mucositis is healed, as well as at weeks 2 and 6 following the end of radiotherapy.

PROJECTED ACCRUAL: A total of 34 patients (17 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of laryngeal cancer with intention to treat by radiotherapy using a 16 fraction 3 week scheme

  * Stage I or II
* No known CNS disease

PATIENT CHARACTERISTICS:

Age:

* 20 to 80

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Hepatic function normal

Renal:

* Renal function normal

Other:

* Not pregnant or nursing
* No serious active infection requiring antibiotic therapy
* No autoimmune disease
* No known seizures
* No psychosocial factors that would preclude study compliance
* No allergies to sargramostim (GM-CSF)
* Willingness to cooperate for regular mirror examination of the larynx

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No concurrent chemotherapy

Endocrine therapy:

* No prior or concurrent corticosteroids
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics

Surgery:

* No major organ allografts

Other:

* No other concurrent investigational drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-10; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.M. Henk, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Trust, London, England, United Kingdom

REFERENCES:
- [Result] McAleese JJ, Bishop KM, A'Hern R, Henk JM. Randomized phase II study of GM-CSF to reduce mucositis caused by accelerated radiotherapy of laryngeal cancer. Br J Radiol. 2006 Jul;79(943):608-13. doi: 10.1259/bjr/55190439. PMID 16823067